CLINICAL TRIAL: NCT01432483
Title: Access Program With Denileukin Diftitox for the Treatment of Patients Currently Receiving Treatment With Commercially Available (Ontak)
Status: No longer available | Type: Expanded Access
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E7272-A001-401
Record Dates: First submitted 2011-09-07; First posted 2011-09-13 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Cancer
Keywords: Cancer; ONTAK; Denileukin diftitox; persistent or recurrent disease; requiring continued delivery of essential cancer therapy
MeSH Terms: conditions — Neoplasms; Recurrence | interventions — denileukin diftitox

INTERVENTIONS:
Drug: Denileukin diftitox (ONTAK) — Given at a dose of 9 or 18mcg/kg/day by intravenous infusion over 30 to 60 minutes for 5 consecutive days every 21 days for 8 cycles.
  Other Names: ONTAK

SUMMARY:
The purpose of this study is to provide continued therapy with Denileukin diftitox (ONTAK) to patients who are currently on therapy and who have no other suitable treatment options, where therapy is requested by their physician.

DETAILED DESCRIPTION:
The Access Program will be provided as long as appropriate according to the judgment of the provider. If Denileukin diftitox (ONTAK) becomes commercially available without restriction, then the access program will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

To receive denileukin diftitox (ONTAK) under this protocol, the patient's physician must request this therapy for the specific patient. Patients may continue treatment with denileukin diftitox if they:

* Are currently on therapy with denileukin diftitox and require ongoing therapy to maintain control of their disease.
* Are willing and able to comply with all aspects of the Access Protocol
* Provide written informed consent to participate

Exclusion Criteria:

Patients are not eligible for the Access Program with denileukin diftitox if they:

• Are not currently on denileukin diftitox therapy

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Gary Palmer, MD, Study Director — Eisai Inc.